# ASSIUT UNIVERSITY HOSPITAL, CLINICAL ONCOLOGY DEPARTMENT

Phase II study of Goserelin for ovarian protection in premenopausal patients receiving cyclophosphamide containing chemotherapy: menstruation outcome.

By:

Ahmed Mohamed Ashraf Saadeldin Abbas 3/17/2018

Phase II study of Goserelin for ovarian protection in premenopausal patients receiving cyclophosphamide containing chemotherapy: menstruation outcome.

### Introduction

The use of adjuvant chemotherapy in younger women with early breast cancer (EBC) has substantially improved the long-term outcome [1]. However, this benefit is associated with long-term toxic effects which are becoming more important as prognosis improves. These include premature menopause and infertility in young pre-menopausal women. The incidence of premature menopause depends on the type and intensity of chemotherapy and the patient's age. In women <35 years old, the long-term (3 years after diagnosis) incidence of amenorrhea is similar to women who have not received chemotherapy, at  $\sim 10\%$ , but this increases to 50% in women between 35 and 40 years old, and can be up to 85% in women >40 years [2]. Premature ovarian failure has major consequences including sexual dysfunction and infertility, and the latter may be of great concern to younger patients with breast cancer and has a bearing in influencing treatment decisions in almost 30% of cases [3].

Currently, there is no standard treatment for preventing chemotherapy-induced ovarian failure. Previous studies have suggested that temporary ovarian suppression with a gonadotropin-releasing hormone (GnRH) analogue may preserve ovarian function both in humans and animal models [4–9]. Clinical data are conflicting. For example, a recent Italian multi-center phase III study

Prevention of Menopause-Induced by Chemotherapy: A Study in Early Breast Cancer Patients-Gruppo Italiano Mamella 6 (PROMISE-GIM6) reported that the use of GnRH analogue, triptorelin during chemotherapy in premenopausal patients with EBC, reduced the occurrence of chemotherapy-induced early menopause with four pregnancies after a 26-month follow-up [one in the chemotherapy alone arm and three in the triptorelin with chemotherapy arm] [10]. In contrast, another trial suggested that the use of goserelin concurrently with neoadjuvant chemotherapy did not significantly reduce incidence of amenorrhea 6 months after the end of chemotherapy compared with those receiving chemotherapy alone and only two pregnancies were recorded [one in each arm] with a follow-up of 2 years [11].

# **Study objectives**

Determination of the role of Goserelin for ovarian protection in premenopausal patients receiving cyclophosphamide containing chemotherapy: menstruation outcome.

#### **Patients and methods**

Eligibility criteria:

- -Premenopausal cancer patients who will recieve Cyclophosphamide-containing chemotherapy.
- -ECOG performance status (PS)  $\leq 2$ .
- -Informed consent will be taken from eligible patients before enrollment

**Exclusion Criteria:** 

Postmenopausal cancer patients

Cancer patients who will receive non Cyclophosphamide containing chemotherapy

# Study design:

This study is a randomized prospective phase II study

Study type: interventional

Study design:

Allocation: randomized

Endpoint classification: efficacy study

Primary endpoint: compare rate of ovarian failure at 1 year between the two treatment groups with ovarian failure defined as the absence of menses in the preceding 6 months and levels of FSH in the postmenopausal range.

Secondary endpoint: median time to recovery of menses from the final dose of goserelin.

Official title: Phase II study of Goserelin for ovarian protection in premenopausal patients receiving cyclophosphamide containing chemotherapy: menstruation outcome.

#### Pretreatment assessment:

Eligible patients will be subjected to the following:

- -History and physical examination especially menstrual history
- -baseline hormonal profile (FSH, LH, E2)

## Treatment protocol:

In this phase II trial, patients will be randomly assigned, in a 1:1 ratio, to standard adjuvant or neoadjuvant chemotherapy with the GnRH agonist goserelin (goserelin group) or to chemotherapy without goserelin (chemotherapy alone group).

For Patients randomly assigned to the goserelin group, goserelin at a dose of 3.6 mg will be administered subcutaneously every 4 weeks beginning 1 week before the initial chemotherapy dose and will be continued to within 2 weeks before or after the final chemotherapy dose.

**Follow up**: All patients will be followed for at least 1 year clinically monthly and by laboratory assessment by hormonal profile (FSH, LH, E2) every 6 months.

## References

- 1. Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Comparisons between different polychemotherapy regimens for early breast cancer: meta-analyses of long-term outcome among 100000 women in 123 randomised trials. Lancet 2012; 379: 432–444.
- 2. Petrek JA, Naughton MJ, Case LD et al. Incidence, time course, and determinants of menstrual bleeding after breast cancer treatment: a prospective study. J ClinOncol 2006; 26: 1045–1051.
- 3. Partridge AH, Gelber S, Peppercorn J et al. Web-based survey of fertility issues in young women with breast cancer. J Clin Oncol 2004; 22: 41744183.
- 4. Ataya K, Rao LV, Lawrence E et al. Luteinizing hormone-releasing hormone agonist inhibits cyclophosphamide-induced ovarian follicular depletion in rhesus monkeys. Biol Reprod 1995; 52: 365–372.
- 5. Blumenfeld Z, Avivi I, Linn S et al. Prevention of irreversible chemotherapy-induced ovarian damage in young women with lymphoma by gonodotrophin-releasing hormone agonist in parallel to chemotherapy. Hum Reprod 1996;
- 11: 1620–1626.6. Blumenfeld Z, Shapiro D, Shteinberg M et al. Preservation of fertility and ovarian function and minimizing gonadotoxicity in young women with systemic lupus erythematosus by chemotherapy. Lupus 2000; 9: 401405.
- 7. Fox K, Ball J, Mick R et al. Preventing chemotherapy-associated amenorrhea (CRA) with leuprolide in young women with early-stage breast cancer. Am Soc Clin Oncol 2001; 20: 25a abstract no. 98.
- 8. Pereya Pacheco B, Mendez Ribas JM, Milone G et al. Use of GnRH analogues for functional protection of the ovary and preservation of fertility during cancer treatment in adolescents: a preliminary report. Gynecol Oncol 2001; 81: 391–397.
- 9. Recchia F, Saggio G et al. Gonadotrophin-releasing hormone analogues added to adjuvant chemotherapy protect ovarian function and improve clinical outcomes in young women with early breast carcinoma. Cancer 2006; 106:514–523.
- 10. Del Mastro L, Boni L, Michelotti A et al. Effect of the gonodotrophin-releasing hormone analogue triptorelin on the occurrence of chemotherapy-induced early menopause in pre-menopausal women with breast cancer. JAMA 2011; 306:269–276.
- 11. Gerber B, von Minckwitz G, Stehle H et al. Effect of luteinizing hormonereleasing hormone agonist on ovarian function after modern adjuvant breast cancer chemotherapy. The GBG 37 ZORO study. J Clin Oncol 2011; 29:2334–2341.